CLINICAL TRIAL: NCT03454126
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled, Single- and Multiple-Ascending Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BIIB095 in Healthy Subjects
Brief Title: Evaluating the Safety, Tolerability, and Pharmacokinetics of BIIB095 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 255HV101; 2017-003982-90 (EudraCT Number)
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteer
Keywords: Chronic pain; Neuropathic pain; Neuralgia; Healthy volunteers
MeSH Terms: conditions — Chronic Pain; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Cohort 1: BIIB095 5 mg (Experimental): Following an overnight fast from food of at least 8 hours, participants will receive a single dose of either BIIB095 5 mg or placebo orally, followed by a fast of at least 4 hours post dose.
  Interventions: Drug: BIIB095; Drug: Placebo
- Cohort 2: BIIB095 25 mg (Experimental): Following an overnight fast from food of at least 8 hours, participants will receive a single dose of either BIIB095 25 mg or placebo orally, followed by a fast of at least 4 hours post dose.
  Interventions: Drug: BIIB095; Drug: Placebo
- Cohort 3: BIIB095 100 mg (Experimental): Following an overnight fast from food of at least 8 hours, participants will receive a single dose of either BIIB095 100 mg or placebo orally, followed by a fast of at least 4 hours post dose.
  Interventions: Drug: BIIB095; Drug: Placebo
- Cohort 4 (Fasted): BIIB095 200 mg (Experimental): Following an overnight fast from food of at least 8 hours, participants will receive a single dose of either BIIB095 200 mg or placebo orally, followed by a fast of at least 4 hours post dose.
  Interventions: Drug: BIIB095; Drug: Placebo
- Cohort 4 (Fed): BIIB095 200 mg (Experimental): After a minimum 2 week washout period, followed by an overnight fast of at least 8 hours, participants will consume a high fat breakfast. Participants will then receive a single dose of either BIIB095 200 mg or placebo orally within 30 minutes after starting the breakfast, followed by a fast from food for at least 4 hours post dose.
  Interventions: Drug: BIIB095; Drug: Placebo
- Cohort 5: BIIB095 400 mg (Experimental): Following an overnight fast from food of at least 8 hours, participants will receive a single dose of either BIIB095 400 mg or placebo orally, followed by a fast of at least 4 hours post dose.
  Interventions: Drug: BIIB095; Drug: Placebo
- Cohort 6: BIIB095 600 mg (Experimental): Following an overnight fast from food of at least 8 hours, participants will receive a single dose of either BIIB095 600 mg or placebo orally, followed by a fast of at least 4 hours post dose.
  Interventions: Drug: BIIB095; Drug: Placebo
- Cohort 7: BIIB095 50 mg BID (Experimental): Participants will receive a single dose of either BIIB095 50 mg or placebo orally BID approximately 12 hours apart from Days 1 to 13, and once in the morning on Day 14. Morning doses will be preceded by an overnight fast from food of at least 8 hours and will be followed by a fast of at least 2 hours post dose. Evening doses will be preceded by a fast from food of at least 2 hours and will be followed by a fast of at least 2 hours post dose.
  Interventions: Drug: BIIB095; Drug: Placebo
- Cohort 8: BIIB095 100 mg BID (Experimental): Participants will receive a single dose of either BIIB095 100 mg or placebo orally BID approximately 12 hours apart from Days 1 to 13, and once in the morning on Day 14. Morning doses will be preceded by an overnight fast from food of at least 8 hours and will be followed by a fast of at least 2 hours post dose. Evening doses will be preceded by a fast from food of at least 2 hours and will be followed by a fast of at least 2 hours post dose.
  Interventions: Drug: BIIB095; Drug: Placebo
- Cohort 9: BIIB095 200 mg BID (Experimental): Participants will receive a single dose of either BIIB095 200 mg or placebo orally BID approximately 12 hours apart from Days 1 to 13, and once in the morning on Day 14. Morning doses will be preceded by an overnight fast from food of at least 8 hours and will be followed by a fast of at least 2 hours post dose. Evening doses will be preceded by a fast from food of at least 2 hours and will be followed by a fast of at least 2 hours post dose.
  Interventions: Drug: BIIB095; Drug: Placebo
- Cohort 10: BIIB095 300 mg BID (Experimental): Participants will receive a single dose of either BIIB095 300 mg or placebo orally BID approximately 12 hours apart from Days 1 to 13, and once in the morning on Day 14. Morning doses will be preceded by an overnight fast from food of at least 8 hours and will be followed by a fast of at least 2 hours post dose. Evening doses will be preceded by a fast from food of at least 2 hours and will be followed by a fast of at least 2 hours post dose.
  Interventions: Drug: BIIB095; Drug: Placebo

INTERVENTIONS:
Drug: BIIB095 — Administered as specified in the treatment arm.
Drug: Placebo — Administered as specified in the treatment arm.

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single- and multiple-ascending oral doses of BIIB095 in healthy participants. The secondary objectives are to characterize the single- and multiple-oral-dose PK of BIIB095 in healthy participants and to investigate the effect of food on the single-oral-dose PK of BIIB095 in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability of the subject to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local subject privacy regulations.
* Must have a body mass index between 18 and 30 kg/m2, inclusive.
* All women of childbearing potential and all men must practice highly effective contraception during the study and for 5 times the half-life or 3 months, whichever is longer, after their last dose of study treatment. In addition, subjects should not donate sperm or eggs during the study and for at least 3 months after their last dose of study treatment.
* Must be in good health as determined by the Investigator, based on medical history and Screening evaluations.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* Significant history of fainting or vaso-vagal attacks, as determined by the Investigator.
* Current condition known to affect cardiac conduction, or a personal or familial history of Brugada syndrome.
* Congenital nonhemolytic hyperbilirubinemia (Gilbert's syndrome).
* History or risk of seizures or a history of epilepsy, significant head injury or related neurological disorders (excluding childhood febrile convulsions), as determined by the Investigator.
* Current enrollment in any other drug, biologic, device, or clinical study, or treatment with an investigational drug or approved therapy for investigational use within 30 days (6 months for biologics) prior to Day -1, or 5 half-lives of the agent, whichever is longer.
* Exposure to more than 4 experimental chemical entities within 12 months prior to the first dosing day.
* Breastfeeding, pregnant, or planning to become pregnant during study participation

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Serious Adverse Events (SAEs) | Signing of Informed Consent (<=28 Days Prior to Day -1, Check-in) to End of Study (Up to 40 Days for Single-Ascending Dose (SAD) Cohorts 1-3 and 5-6; at Least 59 Days for SAD Cohort 4; Up to 53 Days for Multiple-Ascending Dose (MAD) Cohorts 7-10)
  An SAE is any untoward medical occurrence that at any dose:
  Results in death; in the view of the Investigator, places the participant at immediate risk of death (a life threatening event), however, this does not include an event that, had it occurred in a more severe form, might have caused death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; is a medically important event
Percentage of Participants with Adverse Events (AEs) | Signing of Informed Consent (<=28 Days Prior to Day -1, Check-in) to End of Study (Up to 40 Days for Single-Ascending Dose (SAD) Cohorts 1-3 and 5-6; at Least 59 Days for SAD Cohort 4; Up to 53 Days for Multiple-Ascending Dose (MAD) Cohorts 7-10)
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Percentage of Participants with Clinically Significant Abnormalities in Clinical Laboratory Assessments | Signing of Informed Consent (<=28 Days Prior to Day -1, Check-in) to End of Study (Up to 40 Days for Single-Ascending Dose (SAD) Cohorts 1-3 and 5-6; at Least 59 Days for SAD Cohort 4; Up to 53 Days for Multiple-Ascending Dose (MAD) Cohorts 7-10)
Percentage of Participants with Clinically Significant Abnormalities in Vital Signs | Signing of Informed Consent (<=28 Days Prior to Day -1, Check-in) to End of Study (Up to 40 Days for Single-Ascending Dose (SAD) Cohorts 1-3 and 5-6; at Least 59 Days for SAD Cohort 4; Up to 53 Days for Multiple-Ascending Dose (MAD) Cohorts 7-10)
Percentage of Participants with Clinically Significant Abnormalities in 12-Lead Electrocardiogram (ECG) Parameters | Signing of Informed Consent (<=28 Days Prior to Day -1, Check-in) to End of Study (Up to 40 Days for Single-Ascending Dose (SAD) Cohorts 1-3 and 5-6; at Least 59 Days for SAD Cohort 4; Up to 53 Days for Multiple-Ascending Dose (MAD) Cohorts 7-10)
Percentage of Participants with Clinically Significant Abnormalities in Physical Examinations | Signing of Informed Consent (<=28 Days Prior to Day -1, Check-in) to End of Study (Up to 40 Days for Single-Ascending Dose (SAD) Cohorts 1-3 and 5-6; at Least 59 Days for SAD Cohort 4; Up to 53 Days for Multiple-Ascending Dose (MAD) Cohorts 7-10)

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) from Time Zero to the Time of the Last Measurable Concentration (AUClast) | Multiple Time-points on Days 1 through 4 for Single-Ascending Dose (SAD) Cohorts; Multiple Time-points on Days 1 through 15 for Multiple-Ascending Dose (MAD) Cohorts
  Pharmacokinetic (PK) parameter calculated to assess the PK of BIIB095 in blood.
AUC from Time Zero Extrapolated to Infinity (AUC∞) | Multiple Time-points on Days 1 through 4 for Single-Ascending Dose (SAD) Cohorts; Multiple Time-points on Days 1 through 15 for Multiple-Ascending Dose (MAD) Cohorts
  Pharmacokinetic (PK) parameter calculated to assess the PK of BIIB095 in blood.
AUC Within a Dosing Interval (AUCtau) | Multiple Time-points on Days 1 through 4 for Single-Ascending Dose (SAD) Cohorts; Multiple Time-points on Days 1 through 15 for Multiple-Ascending Dose (MAD) Cohorts
  Pharmacokinetic (PK) parameter calculated to assess the PK of BIIB095 in blood.
Maximum Observed Concentration (Cmax) | Multiple Time-points on Days 1 through 4 for Single-Ascending Dose (SAD) Cohorts; Multiple Time-points on Days 1 through 15 for Multiple-Ascending Dose (MAD) Cohorts
  Pharmacokinetic (PK) parameter calculated to assess the PK of BIIB095 in blood.
Trough Concentration (Ctrough) | Multiple Time-points on Days 1 through 4 for Single-Ascending Dose (SAD) Cohorts; Multiple Time-points on Days 1 through 15 for Multiple-Ascending Dose (MAD) Cohorts
  Pharmacokinetic (PK) parameter calculated to assess the PK of BIIB095 in blood.
Time to Cmax (Tmax) | Multiple Time-points on Days 1 through 4 for Single-Ascending Dose (SAD) Cohorts; Multiple Time-points on Days 1 through 15 for Multiple-Ascending Dose (MAD) Cohorts
  Pharmacokinetic (PK) parameter calculated to assess the PK of BIIB095 in blood.
Terminal Elimination Half-Life (t1/2) | Multiple Time-points on Days 1 through 4 for Single-Ascending Dose (SAD) Cohorts; Multiple Time-points on Days 1 through 15 for Multiple-Ascending Dose (MAD) Cohorts
  Pharmacokinetic (PK) parameter calculated to assess the PK of BIIB095 in blood.
Apparent Total Body Clearance (CL/F) | Multiple Time-points on Days 1 through 4 for Single-Ascending Dose (SAD) Cohorts; Multiple Time-points on Days 1 through 15 for Multiple-Ascending Dose (MAD) Cohorts
  Pharmacokinetic (PK) parameter calculated to assess the PK of BIIB095 in blood.
Apparent Volume of Distribution (Vz/F) | Multiple Time-points on Days 1 through 4 for Single-Ascending Dose (SAD) Cohorts; Multiple Time-points on Days 1 through 15 for Multiple-Ascending Dose (MAD) Cohorts
  Pharmacokinetic (PK) parameter calculated to assess the PK of BIIB095 in blood.
Accumulation Ratio (AR) | Multiple Time-points on Days 1 through 4 for Single-Ascending Dose (SAD) Cohorts; Multiple Time-points on Days 1 through 15 for Multiple-Ascending Dose (MAD) Cohorts
  Pharmacokinetic (PK) parameter calculated to assess the PK of BIIB095 in blood.
Amount (Aeu) Excreted in Urine | Multiple Time-points on Days 1 through 4 for Single-Ascending Dose (SAD) Cohorts; Multiple Time-points on Days 1 through 15 for Multiple-Ascending Dose (MAD) Cohorts
  Pharmacokinetic (PK) parameter calculated to assess the PK of BIIB095 in blood.
Percentage (%fe) Excreted in Urine | Multiple Time-points on Days 1 through 4 for Single-Ascending Dose (SAD) Cohorts; Multiple Time-points on Days 1 through 15 for Multiple-Ascending Dose (MAD) Cohorts
  Pharmacokinetic (PK) parameter calculated to assess the PK of BIIB095 in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United Kingdom (2):
  - Research Site, Leeds
  - Hammersmith Medicines Research, London